CLINICAL TRIAL: NCT03139019
Title: Medicaid Incentives for the Prevention of Chronic Diseases: Diabetes Prevention
Acronym: MIPCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: New York State Department of Health (Other Government); Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 818842-1
Record Dates: First submitted 2015-10-12; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Prevention
Keywords: Diabetes prevention; Weight loss; Lifestyle change
MeSH Terms: conditions — Weight Loss | interventions — Microscopy, Electron, Scanning Transmission

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Process incentives (Experimental): Process incentives participants will receive incentives based on visit attendance in the YMCA DPP session. This incentive will be $ 15 for attending each session.
  Interventions: Behavioral: Process incentives
- Outcome incentives (Experimental): Outcome incentives participants will be weighed at 8 and 16 weeks after the program starts and if they have lost 2.5% of their body weight at each time point then they will receive $100 and $140 respectively.
  Interventions: Behavioral: Outcome incentives
- Process and Outcome incentives (Experimental): If assigned to the Process and Outcome arm participants will be informed that they can earn additional incentives for attending DPP classes and losing weight. Participants in this arm can earn $7.50 per DPP class (max 16) and $50 and $70 for achieving 2.5% weight loss at 8 and 16 weeks respectively.
  Interventions: Behavioral: Process and Outcome incentives
- Control arm (No Intervention): If assigned to the Control arm participants will not be eligible for any additional incentives and will just learn the goals of the DPP program itself.

INTERVENTIONS:
Behavioral: Process incentives — Participants will receive cash based incentives for achieving process based measures (class attendance).
  Arms: Process incentives
Behavioral: Outcome incentives — Participants will receive cash based incentives for outcome based measures (weight loss).
  Arms: Outcome incentives
Behavioral: Process and Outcome incentives — Participants will receive cash based incentives for both achieving process based measures (class attendance) and outcome based measures (weight loss).
  Arms: Process and Outcome incentives

SUMMARY:
The relative effectiveness of incentives based on process (e.g. medication adherence) vs. outcome (improvements in blood pressure) is unknown, leading to the key research question: Which approach is more effective? The incentive structure for this initiative is based on best practices in the use of process and outcome measures to address this fundamental question. A series of incentive designs will be conducted to examine the relative effectiveness of equivalent value incentives based on process (e.g. attending smoking cessation counseling sessions), outcomes (e.g. quitting smoking), or a combination of process and outcomes incentives (e.g. attending smoking cessation counseling sessions and quitting smoking). This will also provide an overarching framework for assessing the relative importance of process versus outcome incentives in different contexts and for different populations.

DETAILED DESCRIPTION:
Although great potential exists to promote healthy behaviors through financial incentives, few studies have compared the efficacy and effectiveness of incentives in a Medicaid population. This is important because although financial incentives structured as rewards to individuals substantially improve rates of healthy behaviors, the absolute proportions of people adopting healthier behaviors remain low. Early approaches to financial incentives generally have reflected all-or-nothing thinking by showing that providing incentives is better than not providing incentives, and by assuming that incentives will work similarly across different types of people. But basic research in behavioral economics suggests that how you pay and whom you pay may be critical factors. Furthermore, the relative effectiveness of incentives based on processes vs. outcomes is unknown, and indeed, is one of the most fundamental unresolved questions in the incentive literature. Economists would argue that outcome-based incentives are likely to be more effective because they allow each person to figure out the most efficient path to achieve a desired result. On the other hand, behavioral economists would argue in favor of incentivizing processes because they are simpler and more concrete. Additionally, some ethicists argue that incentivizing processes is fairer because they are effort dependent, and because in some cases the ability to achieve improvements in outcomes may be related to factors people cannot control, such as their environment or their genes. Ultimately, the key question from a health and economic policy standpoint is which approach is more effective. In this regard, improvements in outcomes seem appropriate to incentivize directly because such results are required for incentive programs or other interventions to improve health and/or reduce health care spending. And indeed, there is some limited evidence suggesting that incentives for weight loss, for example, may be more effective than incentives for process measures (eg, attendance) in obesity programs.

The goal of the New York State Medicaid Incentives Plan is to improve clinical outcomes and decrease health expenditures by increasing smoking cessation, lowering high blood pressure, preventing diabetes onset, and enhancing diabetes self-management among Medicaid enrollees in New York State. Several incentive strategies will be explored to promote the use of under-utilized Medicaid benefits and regional resources. The New York State (NYS) Medicaid Incentives Program will target four prevention goals: 1) smoking cessation; 2) lowering high blood pressure; 3) diabetes onset prevention; and 4) diabetes management. For each prevention goal, four treatment arms have been defined. One treatment arm will receive incentives for process activities; one treatment arm will receive incentives for achieving desired outcomes; one treatment arm will receive incentives for both process activities and outcomes; and one arm will serve as a control, receiving no incentives. The smoking cessation incentive program will be piloted in western New York where smoking rates are higher than other regions of the state. Participants will receive direct cash payments for participating in smoking cessation counseling (process), filling nicotine replacement therapy prescriptions (process), and quitting smoking (outcome). 2,332 participants will be recruited for this study. The blood pressure control incentive program will be piloted in New York City where stakeholders are highly engaged and a large population of people at risk for inadequate blood pressure control reside. Participants will receive direct cash payments for attending primary care appointments (process), filling antihypertensive prescriptions (process), and decreasing or maintaining a decreased systolic blood pressure by 10mmHg or achieving another clinically appropriate target (outcome). 488 participants will be recruited for this study. The diabetes management incentive program will be piloted in New York City where the capacity of diabetes self management educators is the greatest. Participants will receive direct cash payment for attending primary care appointments (process), attending diabetes self-management education sessions (process), filling diabetes prescriptions (process), and decreasing their HbA1c by 0.6% or maintaining a level of 8.0% or less (outcome). 660 participants will be recruited for this study. The diabetes onset prevention incentive program will be piloted in western New York and New York City, where the capacity of YMCA Diabetes Prevention Programs is the greatest and well-integrated with stakeholders. Participants will receive lottery tickets for attending YMCA Diabetes Prevention Program sessions (process) and losing or maintaining a reduced weight (outcome). 596 participants will be recruited for this study. Other incentive approaches and research questions will be explored through rapid cycle evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Have been diagnosed as pre-diabetic or high risk for diabetes
* Had a HbA1c test in the last year and if not are willing to get one now
* Medicaid enrolled in NYS

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Process measure: measurement of activities related to diabetes prevention (attending DPP class attendance | During a 16 week program once enrolled
  Number of completed education sessions in a16-week DPP program
Outcome measure: Measure of decrease in weight loss across 16 weeks | During a 16 week period once enrolled
  Weight loss during program.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- NYS Department of Health, Albany, New York, United States

REFERENCES:
- [Background] NYS Medicaid Complete Plan Enrollment, 2010
- [Background] NCQA Patient-Centered Medical Home 2011 Overview. Accessed April 20, 2011. http://www.ncqa.org/tabid/631/default.aspx
- [Background] Office of the Governor Press Release "Governor Cuomo Accepts Recommendations from the Medicaid Redesign Team." February 24, 2011 http://www.governor.ny.gov/press/022411cuomoaccepts_medicaidredesignteam
- [Background] U.S. Census 2010
- [Background] 2010 New York State Managed care Plan Enrollment: A report on managed care enrollment by health plan and county. New York State Department of Health
- [Background] 2009 Medicaid Claims data
- [Background] State Health Facts. Kaiser Family Foundation. Accessed March 28, 2011 http://www.statehealthfacts.org/profileind.jsp?ind=177&cat=4&rgn=34
- [Background] NYS DOH Prevention Quality Indicators. Accessed April 26, 2011. https://apps.nyhealth.gov/statistics/prevention/quality_indicators/start.map;jsessionid=87AA57B85B9BAF52A09F024D8D784077
- [Background] American Legacy Foundation. Saving Lives, Saving Money II: Tobacco-free states spend less on Medicaid. November 2007. Accessed March 28, 2011
- [Background] eQARR Quality Assurance Reporting Requirements New York State. Accessed April 4, 2011. http://www.health.state.ny.us/health_care/managed_care/reports/eqarr/2008/statewide/medicaid/managing_cardiovascular_respiratory_conditions.htm
- [Background] National High Blood Pressure Education Program. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Bethesda (MD): National Heart, Lung, and Blood Institute (US); 2004 Aug. Report No.: 04-5230. Available from http://www.ncbi.nlm.nih.gov/books/NBK9630/ PMID 20821851
- [Background] UnitedHealth Center for Health Reform and Modernization. "The United State of Diabetes: Challenges and opportunities in the decade ahead." Working Paper 5 November 2010.
- [Background] New York State Tobacco Control Program. Leading the way toward a tobacco-free society 2010-2013
- [Background] Centers for Disease Control and Prevention, 2006
- [Background] A guide to the New York State Clean Indoor Air Act. NYS DOH. Access March 28, 2011 http://www.health.state.ny.us/publications/3402/index.htm
- [Background] Centers for Disease Control and Prevention. Behavioral Risk Factor Surveillance System, 2009
- [Background] Heil SH, Higgins ST, Bernstein IM, Solomon LJ, Rogers RE, Thomas CS, Badger GJ, Lynch ME. Effects of voucher-based incentives on abstinence from cigarette smoking and fetal growth among pregnant women. Addiction. 2008 Jun;103(6):1009-18. doi: 10.1111/j.1360-0443.2008.02237.x. PMID 18482424
- [Background] Liu F. Quit attempts and intention to quit cigarette smoking among Medicaid recipients in the USA. Public Health. 2010 Oct;124(10):553-8. doi: 10.1016/j.puhe.2010.05.015. Epub 2010 Sep 15. PMID 20832833
- [Background] McMenamin SB, Halpin HA, Bellows NM. Knowledge of Medicaid coverage and effectiveness of smoking treatments. Am J Prev Med. 2006 Nov;31(5):369-74. doi: 10.1016/j.amepre.2006.07.015. Epub 2006 Sep 25. PMID 17046407
- [Background] Centers for Disease Control and Prevention. Leading Causes of Deaths. Accessed March 29, 2011 http://www.cdc.gov/nchs/fastats/lcod.htm
- [Background] NYS (county level) Data Source: NYS Department of Health, Expanded Behavioral Risk Factor Surveillance System (Expanded BRFSS), http://www.nyhealth.gov/statistics/brfss/expanded/. 2008-2009
- [Background] Elzubier AG, Husain AA, Suleiman IA, Hamid ZA. Drug compliance among hypertensive patients in Kassala, eastern Sudan. East Mediterr Health J. 2000 Jan;6(1):100-5. PMID 11370321
- [Background] Shaya FT, Du D, Gbarayor CM, Frech-Tamas F, Lau H, Weir MR. Predictors of compliance with antihypertensive therapy in a high-risk medicaid population. J Natl Med Assoc. 2009 Jan;101(1):34-9. doi: 10.1016/s0027-9684(15)30808-7. PMID 19245070
- [Background] Ormond BA, Spillman BC, Waidmann TA, Caswell KJ, Tereshchenko B. Potential national and state medical care savings from primary disease prevention. Am J Public Health. 2011 Jan;101(1):157-64. doi: 10.2105/AJPH.2009.182287. Epub 2010 Nov 18. PMID 21088270
- [Background] National Diabetes Information Clearing House Accessed March 30, 2011 http://diabetes.niddk.nih.gov/dm/pubs/statistics/#dud
- [Background] U.S. Preventive Services Task Force. The Guide to Clinical Preventive Services 2010 - 2011: Recommendations of the U.S. Preventive Services Task Force. Rockville (MD): Agency for Healthcare Research and Quality (US); 2010 Aug. Report No.: 10-05145. Available from http://www.ncbi.nlm.nih.gov/books/NBK56707/ PMID 21850778
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Hamman RF, Wing RR, Edelstein SL, Lachin JM, Bray GA, Delahanty L, Hoskin M, Kriska AM, Mayer-Davis EJ, Pi-Sunyer X, Regensteiner J, Venditti B, Wylie-Rosett J. Effect of weight loss with lifestyle intervention on risk of diabetes. Diabetes Care. 2006 Sep;29(9):2102-7. doi: 10.2337/dc06-0560. PMID 16936160
- [Background] Ackermann RT, Finch EA, Brizendine E, Zhou H, Marrero DG. Translating the Diabetes Prevention Program into the community. The DEPLOY Pilot Study. Am J Prev Med. 2008 Oct;35(4):357-63. doi: 10.1016/j.amepre.2008.06.035. PMID 18779029
- [Background] Amundson HA, Butcher MK, Gohdes D, Hall TO, Harwell TS, Helgerson SD, Vanderwood KK; Montana Cardiovascular Disease and Diabetes Prevention Program Workgroup. Translating the diabetes prevention program into practice in the general community: findings from the Montana Cardiovascular Disease and Diabetes Prevention Program. Diabetes Educ. 2009 Mar-Apr;35(2):209-10, 213-4, 216-20 passim. doi: 10.1177/0145721709333269. PMID 19321807
- [Background] Sjostrom CD, Lissner L, Wedel H, Sjostrom L. Reduction in incidence of diabetes, hypertension and lipid disturbances after intentional weight loss induced by bariatric surgery: the SOS Intervention Study. Obes Res. 1999 Sep;7(5):477-84. doi: 10.1002/j.1550-8528.1999.tb00436.x. PMID 10509605
- [Background] Volpp KG, Loewenstein G, Troxel AB, Doshi J, Price M, Laskin M, Kimmel SE. A test of financial incentives to improve warfarin adherence. BMC Health Serv Res. 2008 Dec 23;8:272. doi: 10.1186/1472-6963-8-272. PMID 19102784
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] Volpp KG, Pauly MV, Loewenstein G, Bangsberg D. P4P4P: an agenda for research on pay-for-performance for patients. Health Aff (Millwood). 2009 Jan-Feb;28(1):206-14. doi: 10.1377/hlthaff.28.1.206. PMID 19124872
- [Background] Balamurugan A, Ohsfeldt R, Hughes T, Phillips M. Diabetes self-management education program for Medicaid recipients: a continuous quality improvement process. Diabetes Educ. 2006 Nov-Dec;32(6):893-900. doi: 10.1177/0145721706294787. PMID 17102156
- [Background] Norris SL, Engelgau MM, Narayan KM. Effectiveness of self-management training in type 2 diabetes: a systematic review of randomized controlled trials. Diabetes Care. 2001 Mar;24(3):561-87. doi: 10.2337/diacare.24.3.561. PMID 11289485
- [Derived] Chin JY, Matson J, McCauley S, Anarella J, Gesten F, Roohan P. The impact of financial incentives on utilization and outcomes of diabetes prevention programs among Medicaid managed care adults in New York state. Contemp Clin Trials. 2020 Apr;91:105960. doi: 10.1016/j.cct.2020.105960. Epub 2020 Feb 19. PMID 32087338